CLINICAL TRIAL: NCT01927770
Title: Randomized Trial of Consent Interventions for NIH Whole Exome and Whole Genome Sequencing Studies
Brief Title: A Study of Consent Forms for Whole Exome and Whole Genome Sequencing
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130171; 13-HG-0171
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Whole Genome Sequencing
Keywords: WES; Informed Consent; WGS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- WES/WGS: Eligible adults (or parents of eligible children) consenting to enroll in an NIH study thatincludes WES/WGS.

SUMMARY:
Background:

The purpose of this study is to investigate the process of consenting participants to whole exome/genome sequencing and its outcomes. It is unknown how best to consent people to this new technology. NO GENOME SEQUENCING IS OFFERED AS PART OF THIS STUDY. This protocol is a companion to other NIH studies that involve genomic sequencing. Participants must be enrolled in a parent NIH study that is collaborating on this consent study to be eligible. Currently this involves only one NIH study.

Objectives:

- To learn the best way to help participants understand sequencing, so they can decide whether to join studies that use it.

Eligibility:

* Adults at least 18 years old who are enrolled in a National Institutes of Health (NIH) study that uses WES/WGS.
* Adults at least 18 years old whose children are enrolled in an NIH study that uses WES/WGS.

Design:

* Participants will take part in the study either in person or over the phone.
* Participants will review two sequencing consent forms with a genetic counselor.
* Before and after meeting with the counselor, participants will answer several questions about sequencing. Each questionnaire will take about 15 minutes.
* Six weeks later, participants will answer questions about sequencing. This will take about 15 minutes.

DETAILED DESCRIPTION:
Consent to participant in studies that include whole exome and whole genome sequencing (WES/WGS) studies and to receive results present challenges to achieving informed consent due to the scope, depth and uncertainty of the information. NIH Intramural studies increasingly involve WES/WGS to identify elusive primary variants. This umbrella protocol aims to compare an evidence-based consent for WES/WGS to a standard consent in collaboration with ongoing and future NIH studies. An equivocal hypothesis will be tested to evaluate whether informed choice and perceptions of uncertainty differ between two consent

groups. A mixed-methods design is proposed that starts with a qualitative mental-model pilot

study to revise an expert opinion consent intervention by integrating lay-person response

preferences. Following development of this evidence-based intervention, a randomized two- factor design will be used for a quantitative survey study conducted in conjunction with a

number of NIH studies conducting WES/WGS to test for differences between two consent

models. A descriptive analysis of the audiotaped consent process will also be conducted to

assess differences in the content or extent of the process, and related outcomes of satisfaction and decisional conflict will also be assessed.

ELIGIBILITY:
* INCLUSION CRITERIA:

Eligible adults (greater than or equal to 18 years of age) consenting to enroll in an NIH study that includes WES/WGS. Parents of eligible children (<18 years of age) consenting to enroll their child(ren) in an NIH study that includes WES/WGS. Participants must be cognitively able to consent and fluent in written and spoken English.

EXCLUSION CRITERIA:

Children (<18 years of age). Non-English speaking participants (until the study has evolved to be able to use translations of the interventions into Spanish).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents and eligible children.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2016-03-07 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
A | Ongoing
  To contrast the efficacy of an evidence-based streamlined consent model (based upon the integration of an expert opinion model and laypersons responses using a mental- models approach) to a standard NIH consent in consenting adult and parent participants to undergo WES/WGS within NIH Intramural studies.
B | Ongoing
  To quantitatively assess changes in understanding, perceptions of uncertainty and informed choice between the two consent interventions, assuming equivalency.
C | Ongoing
  To describe satisfaction,decisional conflict and residual questions and concerns following use of each consent intervention.
D | Ongoing
  To compare the content, dialogue and time spent in the consent discussions between interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Sapp, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ayuso C, Millan JM, Mancheno M, Dal-Re R. Informed consent for whole-genome sequencing studies in the clinical setting. Proposed recommendations on essential content and process. Eur J Hum Genet. 2013 Oct;21(10):1054-9. doi: 10.1038/ejhg.2012.297. Epub 2013 Jan 16. PMID 23321621
- [Background] Biesecker LG, Mullikin JC, Facio FM, Turner C, Cherukuri PF, Blakesley RW, Bouffard GG, Chines PS, Cruz P, Hansen NF, Teer JK, Maskeri B, Young AC; NISC Comparative Sequencing Program; Manolio TA, Wilson AF, Finkel T, Hwang P, Arai A, Remaley AT, Sachdev V, Shamburek R, Cannon RO, Green ED. The ClinSeq Project: piloting large-scale genome sequencing for research in genomic medicine. Genome Res. 2009 Sep;19(9):1665-74. doi: 10.1101/gr.092841.109. Epub 2009 Jul 14. PMID 19602640
- [Background] Dormandy E, Michie S, Hooper R, Marteau TM. Low uptake of prenatal screening for Down syndrome in minority ethnic groups and socially deprived groups: a reflection of women's attitudes or a failure to facilitate informed choices? Int J Epidemiol. 2005 Apr;34(2):346-52. doi: 10.1093/ije/dyi021. Epub 2005 Feb 28. PMID 15737971
- [Derived] Turbitt E, Chrysostomou PP, Peay HL, Heidlebaugh AR, Nelson LM, Biesecker BB. A randomized controlled study of a consent intervention for participating in an NIH genome sequencing study. Eur J Hum Genet. 2018 May;26(5):622-630. doi: 10.1038/s41431-018-0105-7. Epub 2018 Feb 16. PMID 29453419
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-HG-0171.html